CLINICAL TRIAL: NCT06092203
Title: Assessment of Health-Related Quality of Life for Pediatric Patients With Urinary Stone Disease.
Brief Title: Quality of Life for Pediatric Urolithiasis
Acronym: Elattar
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed R. EL-Nahas, Professor of Urology, Mansoura University
Other Study IDs: 2278
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Pediatric ALL
Keywords: Urolithiasis; Quality of life; PCNL; SWL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Urolithiasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Pediatric patients who underwent treatment for utrollithiasis.
- Control: Cross-matched group of healthy children.

SUMMARY:
The aim of this study is to assess the quality of life (QoL) in pediatric patients with urinary stone disease.

DETAILED DESCRIPTION:
This study will assess the quality of life (QoL) in pediatric patients with urinary stone disease using the pediatric quality of life (PedsQol) questionnaire in comparison to normal healthy age/sex matched population.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had urinary stones

Exclusion Criteria:

1. Patients presenting with obstructive uropathy or urosepsis.
2. Recent (less than 4 weeks) surgical intervention for urinary stone disease.
3. Indwelling urinary catheters or stents (urethral catheter, ureteral stents or nephrostomy tube).
4. Associated mental illness or cognitive dysfunction.
5. Associated chronic medical illness that may compromise QoL.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All pediatric patients with urolithiasis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
The PedsQL questionnaire | 12 months
  comparison of overall PedsQL score between pediatric urolithiasis patients and normal healthy age/sex matched population.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed R EL-Nahas, MD, Principal Investigator — Mansoura University
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No